CLINICAL TRIAL: NCT02822378
Title: Randomized Control Trial of Dietary Supplementation With Dried Plums on Bone Density, Geometry and Estimated Bone Strength in Postmenopausal Women
Brief Title: Dried Plums and Bone Health in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: California Dried Plum Board (Other)
Responsible Party: Principal Investigator, Mary Jane DeSouza, Professor of Kinesiology and Physiology, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Study00004252
Record Dates: First submitted 2016-05-27; First posted 2016-07-04 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal Osteoporosis; Human; Female; Non-pharmacologic therapy
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ca2+/VitD Control (Experimental): Participants will take calcium and vitamin D supplements for the duration of the baseline and intervention. Participants will be asked to refrain from consumption of dried plums for the duration of the intervention (52 weeks).
  Interventions: Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D supplement
- 50g Dried Plums (Experimental): Participants will take calcium and vitamin D supplements for the duration of the baseline and intervention. Additionally, participants will be provided with dried plums and asked to consume 6 (50g) dried plums per day for the duration of the intervention (52 weeks).
  Interventions: Dietary Supplement: Dried Plum; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D supplement
- 100g Dried Plums (Experimental): Participants will take calcium and vitamin D supplements for the duration of the baseline and intervention. Additionally, participants will be provided with dried plums and asked to consume 12 (100g) dried plums per day for the duration of the intervention (52 weeks).
  Interventions: Dietary Supplement: Dried Plum; Dietary Supplement: Calcium supplement; Dietary Supplement: Vitamin D supplement

INTERVENTIONS:
Dietary Supplement: Dried Plum — Participants randomized to the 50g dried plum group will consume 6 dried plums per day for the duration of the 52 week intervention. Participants randomized to the 100g dried plum group will consume 12 dried plums per day for the duration of the 52 week intervention.
  Other Names: Prunes
  Arms: 100g Dried Plums; 50g Dried Plums
Dietary Supplement: Calcium supplement — All participants will consume calcium supplements for the duration of baseline and intervention.
Dietary Supplement: Vitamin D supplement — All participants will consume vitamin D supplements for the duration of baseline and intervention.

SUMMARY:
Postmenopausal women often seek non-pharmacologic interventions for the protection of bone health. Previous research in humans and rodents has indicated that dietary dried plum consumption may be beneficial for bone health, especially in postmenopausal women. However, it is unknown in what quantity dried plums need to be consumed to be of benefit and through what mechanisms dried plums act to impact bone health. Therefore, the purpose of this study is to evaluate the impact of 52 weeks of dried plums consumption in varying quantities on bone mineral density (BMD), bone geometry, and estimated bone strength in postmenopausal women. The investigators also seek to evaluate the mechanisms underlying the effects of dried plums as a dietary supplement by assessing polyphenols and the bioavailable conjugated metabolites in the urine of postmenopausal women taking different doses of dietary dried plums. The investigators aim to further investigate the mechanisms of dried plum action on bone by measuring markers of bone metabolism in response to dried plum consumption.

DETAILED DESCRIPTION:
Given the current high incidence of osteoporosis, reducing the risk of osteoporosis development is essential. Recent estimates, based on the 2010 US Census, indicate that approximately 10.3 million people age 50 and older have osteoporosis. By 2030 the prevalence of osteoporosis for women 50 years and older is projected to reach 13.6 million. Postmenopausal osteoporosis is characterized not only by hypoestrogenism, but also by increased production of reactive oxygen species, oxidative stress, and inflammatory response. Current first line strategies are treatment of osteoporosis with pharmacologic approaches. Complementary recommendations include the maintenance of calcium (Ca2+) and vitamin D (VitD) intake to meet the current recommendations. Although the anti-resorptive therapies are effective they are also associated with an array of negative side effects, which reduce patient compliance to use of the therapy.

Non-pharmacologic options to reducing the risk of bone loss are becoming more attractive to many postmenopausal women. The phenolics and bioavailable conjugated metabolites found in dried plums are proposed to modulate the inflammatory signaling pathways and have the potential to influence bone formation and bone resorption, thus modulating the risk of bone loss. The investigators are conducting a 52 week dose ranging randomized controlled trial that builds upon previous rodent and human work and addresses the experimental design limitations of the previous work, to assess bone outcomes with clinical (BMD) and mechanistic (bone geometry, bone metabolism markers, and inflammation markers) techniques. Additionally, this study will include a detailed assessment of the phenolics in the dried plums to explore the relationship between these compounds and bone outcomes.

Participants will participate in a 1-2 week screening period followed by a 1-2 week baseline period. At the end of baseline randomization to 1 of 3 groups will occur (Ca2+ and VitD only; 50g Dried Plums/day and Ca2+ and VitD; 100g Dried Plums/day and Ca2+ and VitD). Dried plums and Calcium/Vitamin D supplements will be provided to participants for the duration of the intervention. At the beginning of the 52 week intervention participants will begin consumption of dried plums and will be given a run in period where the number of dried plums consumed per day increases slowly to minimize the side effects felt by the participants. The dried plums will be consumed as snacks in the morning, midday, and in the evening. Participants will visit the laboratory for testing every 4 weeks during the 52 week intervention, with more testing occurring during weeks 12, 24, 36, and 52 than the other testing periods.

At testing period visits participants will be asked to complete some or all of the following: body weight measurement; blood sampling; 24-hour urine collection; stool sample collection; DXA scan; peripheral quantitative computed tomography (pQCT) scan; completion of health, physical activity, and nutrition questionnaires; completion of supplement/symptom, diet, and physical activity logs.

A total of 300 participants will be enrolled and screed with an expected randomization of 79 participants per group. The investigators anticipate a 20% drop-out rate between baseline and week 52, thus will anticipate having a final sample size of 63 participants per group complete the study. This sample size provides over 80% power to detect differences with the primary BMD, bone geometry, and bone strength variables.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women
* not severely obese (BMI < 40 kg/m2);
* healthy (determined by a screening questionnaire, complete metabolic panel);
* willing to include dried plums in their daily diet;
* not taking any natural dietary supplement containing phenolics, blueberries or apples for at least 2 months prior to study entry; can stop for 2 months to meet entry criteria
* non-smoking; ambulatory;
* low BMD as measured by dual energy X-ray absorptiometry (DXA). Eligible BMD values (T-scores) for DXA measures of the lumbar spine, total hip and/or femoral neck will correspond to T-scores between 0 and -3.0.

Exclusion Criteria:

* Women who regularly consume dried plums, dried apples, prune juice, or heavy consumers of blueberries (1 cup or more/day). Potential volunteers who will refrain from consumption of the afore mentioned foods for the duration of the study will become eligible after a 2 month washout period;
* vitamin D deficiency (<20 ng/mL);
* history of vertebral fracture or fragility fracture of the wrist, humerus, hip or pelvis after age 50 yr);
* untreated hyper- or hypothyroidism;
* current hyper- or hypoparathyroidism;
* significantly impaired renal function; high potassium
* current hypo- or hypercalcemia;
* history of spinal stenosis;
* history of heart attack, stroke, thromboembolism, kidney disease, malabsorption syndrome, seizure disorders;
* positive for HIV, Hep-C or Hep-B surface antigen and malignancy.
* Use of the following agents affecting bone metabolism:

  * intravenous bisphosphonates at any time;
  * fluoride (for osteoporosis) within the past 24 months;
  * denosumab at any time;
  * bisphosphonates, parathyroid hormone or strontium within the past 12 months;
  * calcitonin or selective estrogen receptor modulators within the past 12 months;
  * systemic oral or transdermal estrogen within the past 3 months;
  * systemic glucocorticosteroids (≥ 5 mg prednisone equivalent per day for more than 10 days); or
  * tibolone within the past 3 months.
* Participants who will not consume study therapy or will not stop taking natural product supplements of their own selection.

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2016-06-01; Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in areal bone mineral density (via DXA) of the lumbar spine, total hip, and femoral neck | at screening, week 24, and week 52
  Percent change in areal BMD measured during screening, and weeks 24 and 52 of the 52 week dietary intervention at the lumbar spine, total hip, and femoral neck.

SECONDARY OUTCOMES:
Percent change from baseline in DXA hip structural analysis | at screening, week 24, and week 52
  Percent change in hip structural analysis (HSA) measured during screening, and weeks 24 and 52 of the 52 week dietary intervention at the total hip.
Percent change from baseline in DXA spine trabecular bone score | at screening, week 24, and week 52
  Percent change in trabecular bone score (TBS) measured during screening, and weeks 24 and 52 of the 52 week dietary intervention at the lumbar spine.
Percent change from baseline in pQCT volumetric BMD of the tibia and radius | at baseline, week 24, and week 52
  Percent change in volumetric BMD, cortical and trabecular compartments, measured during baseline, and weeks 24 and 52 of the 52 week dietary intervention at the tibia and radius. The combination of measurements will provide an overall picture of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in pQCT geometry measurements of the tibia and radius | at baseline, week 24, and week 52
  Percent change in bone geometry estimates measured during baseline, and weeks 24 and 52 of the 52 week dietary intervention at the tibia and radius. The combination of measurements will provide an overall picture of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Percent change from baseline in pQCT strength measurements of the tibia and radius | at baseline, week 24, and week 52
  Percent change in bone strength estimates measured during baseline, and weeks 24 and 52 of the 52 week dietary intervention at the tibia and radius. The combination of measurements will provide an overall picture of the 3-dimensional structure of a weight bearing (tibia) and non-weight bearing (radius) site and how the sites are impacted by the intervention.
Change from baseline in bone turnover markers | at baseline, week 12, week 24, week 36, and week 52
  Change in serially-sampled fasting serum concentrations of bone formation (N-terminal type 1 procollagen; P1NP) and bone resorption (crosslaps; CTx) before, during and after the dietary intervention. The combined measures will provide information regarding changes in the rate of bone resorption and bone formation.

OTHER OUTCOMES:
Change from baseline in cellular bone metabolism | at baseline, week 12, week 24, week 36, and week 52
  Change in serially-sampled fasting serum concentrations of bone signaling markers (i.e., Insulin like growth factor-1 [IGF-1], osteoprotegerin [OPG], receptor activator of nuclear factor kappaB ligand [RANKL], and sclerostin [SOST]) before, during and after the dietary intervention. Changes in these variables will assist in understanding the underlying mechanisms behind changes in the rates of bone resorption and bone formation.
Change from baseline in urine phenolic concentrations | at baseline and every 4 weeks during the intervention
  Change in serially-sampled 24 hour urine concentrations of phenolic compounds attributable to dried plum consumption.
Change from baseline in serum phenolic concentrations | at baseline, week 12, week 24, week 36, and week 52
  Change in serially-sampled fasting serum concentrations of phenolic compounds attributable to dried plum consumption.
Change from baseline in expression of inflammatory markers | at baseline, week 12, week 24, week 36, and week 52
  Change in peripheral blood mononuclear cell (PBMC) gene expression of inflammatory markers before, during and after the dietary intervention. Additionally, the relationship between the changes in gene expression of inflammation markers and bone outcomes will be explored. The combined changes of the gene expression of inflammatory markers will provide a comprehensive picture of the inflammatory environment of the participants before, during and following the dietary intervention. This comprehensive picture will assist in understanding the mechanisms by which the inflammatory environment contributes to bone loss in postmenopausal women and how the dietary intervention impacts these factors.
Change from baseline in gut microbiome | at baseline, week 24, and week 52
  Serially-sampled stool samples for assessment of changes in the gut microbiome before, during and after the dietary intervention. Additionally, the relationship between the changes in the gut microbiome and bone outcomes will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jane De Souza, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- Women's Health and Exercise Laboratories, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Damani JJ, Rogers CJ, Lee H, Strock NC, Koltun KJ, Williams NI, Weaver C, Ferruzzi MG, Nakatsu CH, De Souza MJ. Effects of Prune (Dried Plum) Supplementation on Cardiometabolic Health in Postmenopausal Women: An Ancillary Analysis of a 12-Month Randomized Controlled Trial, The Prune Study. J Nutr. 2024 May;154(5):1604-1618. doi: 10.1016/j.tjnut.2024.03.012. Epub 2024 Mar 13. PMID 38490532
- [Derived] Damani JJ, Oh ES, De Souza MJ, Strock NC, Williams NI, Nakatsu CH, Lee H, Weaver C, Rogers CJ. Prune Consumption Attenuates Proinflammatory Cytokine Secretion and Alters Monocyte Activation in Postmenopausal Women: Secondary Outcome Analysis of a 12-Mo Randomized Controlled Trial: The Prune Study. J Nutr. 2024 May;154(5):1699-1710. doi: 10.1016/j.tjnut.2023.11.014. Epub 2023 Nov 19. PMID 37984741
- [Derived] De Souza MJ, Strock NCA, Williams NI, Lee H, Koltun KJ, Rogers C, Ferruzzi MG, Nakatsu CH, Weaver C. Prunes preserve hip bone mineral density in a 12-month randomized controlled trial in postmenopausal women: the Prune Study. Am J Clin Nutr. 2022 Oct 6;116(4):897-910. doi: 10.1093/ajcn/nqac189. PMID 35798020